CLINICAL TRIAL: NCT01769092
Title: Double Blind Placebo Controlled Trial of Anticonvulsant Effects of n-3 PUFAs in Human Subjects With Epilepsy
Brief Title: Clinical Trial of the Effects of DHA in the Treatment of Seizure Disorders
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: North York General Hospital (Other); Ontario Brain Institute (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCNM1302
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy (Treatment Refractory)
Keywords: Epilepsy; Seizure; Fish Oil
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Fish Oils; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish Oil (Experimental): Each capsule contains 625 mg of fish oil (100 mg EPA & 250 mg DHA). Participants will take 12 capsules per day over 6 months.
  Interventions: Dietary Supplement: Fish Oil
- Safflower Oil (Placebo Comparator): Each capsule will contain 625 mg of Safflower oil. Participants will take 12 capsules per day over 6 months.
  Interventions: Other: Safflower Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — The daily dose is divided; capsules are taken with meals for a period of 6 months.
  Other Names: Docosahexanoic acid; EPA
  Arms: Fish Oil
Other: Safflower Oil — Daily dose of safflower oil taken in divided doses as capsules and consumed with meals.
  Arms: Safflower Oil

SUMMARY:
For many years, there has been interest in the question of whether a special diet of some sort could be used to help control epileptic seizures. The ketogenic diet has been used since the 1920s, but it is used only in children, and is nutritionally unbalanced. It is typically withdrawn after 3 years. The ketogenic diet unfortunately, offers no long-term solution to seizure control.

Our preliminary research now suggests that there may be a healthy, long-term dietary approach to controlling seizures.

Based on our animal work and published clinical studies the investigators hypothesize that a DHA dose of 3 g/day will reduce seizure frequency in patients with intractable seizures.

DETAILED DESCRIPTION:
This will be a small, double-blind study involving placebo and 3 g/day of DHA. There will be a one-month baseline period, followed by a six month treatment period.

1. Neurologists from the North York General Hospital or Toronto Western Hospital will refer patients being treated for intractable epilepsy.
2. Patients will be contacted by phone by the study coordinator, who will explain the study and ask about willingness to participate. Inclusion and exclusion criteria will be discussed, as well as the patient's responsibilities. It will be made clear that there will be no cost to the patient.
3. If patients are interested, a letter will be sent to them. The letter will contain a description of the study, the patient's responsibilities if he/she agrees to participate, and an explanation of informed consent.
4. One week after the letter, the study coordinator will again contact the patients by phone, answer any questions, and

   - if the patient is willing to participate - set up the initial visit.
5. At the initial visit, the study coordinator will give the subject written and verbal information. Patients will be asked to sign an informed consent form. They will be given a seizure diary, to keep during the first month (prior to treatment) and to continue for the six months of treatment. The diary will record the frequency/type of seizures.

   The study physician will review the medial history (seizure frequency/type), medications and blood work to be taken to measure serum levels of AEDs and n-3 PUFAs. About two teaspoons of extra blood will be taken and stored for possible future assays.

   The study coordinator will then provide the patients with their appropriate capsules for the first three months of the trial. The rest will be mailed. The patient will receive written instructions on how to take the capsules. Only the study coordinator will know the patients' group assignments. (A sealed back-up of the code will be left with Dr. Burnham.) Patients will be given the study coordinator's cell phone number with instructions to call if they feel unwell at any time. If serious problems occur, the study coordinator will refer patients to the Emergency Department.
6. Weekly telephone calls: Participants will receive scheduled weekly telephone calls from the study coordinator to collect any information recorded in the seizure diaries during the one month baseline period continuing through the sixth month treatment period.
7. After the last month of the trial, a second in-person visit will be scheduled to re-examine the patient, and order more blood work. (Two teaspoons of the blood will be reserved for possible future assays.) At the end of the visit, The study coordinator will debrief the patient and give him/her a letter of thanks from the P.I. The patient will then be told where he/she can purchase DHA if he/she wants to continue.
8. Data will be analyzed by Dr. Burnham. After data analysis, patients will be informed about the results of the whole by letter.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older
* Female subjects must be using a form of contraception
* >1 seizures per month
* EEG confirmation of seizure activity (no non-epileptic seizures)
* Agrees to comply with study procedures, and keep seizure diary
* Agrees not to make any major deviations from current diet (especially fish intake) or medications (type, dosage)
* Agrees to having portions of blood samples stored for assays
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Use of significant amounts of fish oil or flax oil (omega-3) supplements within 8 weeks of the study.
* Allergy or sensitivity to fish, fish oil, coconut oil, olive oil, hemp oil, safflower oil, flax seed oil, or soybean oil
* Cognitive impairment (I.Q. below 70) and/or inability to give informed consent.
* Failure to understand English
* Subjects taking regular warfarin or aspirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Seizure Diary | 6 months
  The primary outcome measure of the study will be a measure of the number of seizures each month as recorded in a seizure diary - a record kept under the supervision of the study coordinator.

SECONDARY OUTCOMES:
Serum poly-unsaturated fatty acid levels | 6 months
  Blood samples will be banked to allow for an assessment of change in blood levels of poly-unsaturated fatty acids between baseline and final study visit (6 months)
Serum anticonvulsant levels | 6 months
  Blood samples will be assessed for levels of anti-convulsant medications at baseline and 6 month time periods
Adverse reactions | 6 months
  All adverse reactions incurred by all participants within the study will be collected, reported and assessed by type, intensity, severity, duration, and relationship to the study products

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Hwang, MD, Principal Investigator — North York General Hospital; Mac Burnham, PhD, Study Director — University of Toronto Epilepsy Research Program (UTERP); Peter Carlen, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Findings will be shared with participants upon request. Results will be disseminated at epilepsy conferences.